CLINICAL TRIAL: NCT02711865
Title: Predictive Biomarkers for IGF1R Targeted Therapy in Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-54-15
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumors that will be removed from women operated on for ovarian cancer.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MK-0646: Tumor specimens removed from 20 women with ovarian cancer are injected into 40 mice treated with the IGF1R antibody MK-0646. The drug will be administered twice weekly, via IP injection at a dose of 500 microgram per animal.
  Interventions: Biological: IGF1R antibody MK0646
- Control: Tumor specimens removed from 20 women with ovarian cancer are injected into 40 mice who receive no other treatment.
  Interventions: Other: Saline solution

INTERVENTIONS:
Biological: IGF1R antibody MK0646
  Groups: MK-0646
Other: Saline solution
  Groups: Control

SUMMARY:
The main goal of this study is to employ a novel proteomic approach to identify predictive tumor biomarkers that will increase the efficacy of insulin-like growth factor (IGF1R) targeted therapy in epithelial ovarian cancer. It is expected that these predictive biomarkers will be applied to increase the response rate in selected groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian cancer

Exclusion Criteria:

* All others

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty fresh ovarian cancer specimens will be obtained from patients operated on and treated at the Hillel Yaffe Medical Center.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Responsive to IGF1R therapy | One year
  Mean tumor volume will be calculated and growth inhibition will be reported as the percentage decrease of tumor volume compared with the control.

SECONDARY OUTCOMES:
Proteomic Signature of IGF1R Responsive Tumors | One year
  Mass Spectrometry will be used to compare IGF1R responsive and non-responsive tumors to identify the proteins associated with sensitivity to IGF1R therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Bruchim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No